CLINICAL TRIAL: NCT04678726
Title: Nurse-performed Lung Ultrasound Versus Chest Radiography for Detection of Pneumothorax After Mediastinal Drainage Removal Post Cardiac Surgery.
Brief Title: Nurse-performed Lung Ultrasound Versus Chest Radiography for Detection of Pneumothorax.
Status: Withdrawn | Type: Observational
Why Stopped: COVID interference in the ability to initiate the study.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 17-6203
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2022-11

CONDITIONS: Pneumothorax; Cardiac Surgery
Keywords: Chest tube removal
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung ultrasound assessment for ruling out pneumothorax — Patients who have undergone heart surgery and have decided to enroll in our study, will have the standard chest x-ray and an additional lung ultrasound. Within a maximum of two hours of the chest tube removal, the standard chest x-ray will be performed, and then a different nurse will perform the lung ultrasound to check for pneumothorax.
  Other Names: Portable chest x-ray

SUMMARY:
This is a prospective, single-center, observational, cross-sectional cohort study, comparing nurse-performed bedside lung ultrasound to standard portable CXR, for the detection of pneumothorax in the cardiac surgery patient population, following chest tube removal. This study aims to be conducted at an academic, tertiary adult center cardio-vascular intensive care unit (CVICU at TGH).

DETAILED DESCRIPTION:
To avoid the accumulation of blood and fluids in the mediastinum or pleural cavities after cardiac surgery, mediastinal and pleural drains are routinely used. The rate of pneumothorax following chest drain removal is approximately 1.5-13%, resulting in increased patient morbidity and hospital stay. The standard method for the determination of pneumothorax (PNX) in most institutions is to obtain a chest radiography (CXR) following chest tube removal, but the reliability of the supine anteroposterior chest radiography is not utter, with up to 30% of pneumothoraxes misdiagnosis. The delay of ordering, performing and interpreting a CXR post mediastinal tube removal, results in potential delay in patients transfers, with an estimated cost savings of omitting an additional chest radiography, of approximately $10 000 per year.

Lung ultrasound (LUS) is recommended for detection of pneumothorax as per evidence-based guidelines and expert consensus. Lung ultrasound is a safe technique due to minimal radiation, with the potential for immediate results when compared with the standard CXR. LUS has high accuracy for PNX detection, with better pooled sensitivities (78.6%) when compared to CXR (39.8%) and equal specificity (98.4 vs 99.3%). In intensive care units, those results have been reproducible, with LUS having greater sensitivity than CXR for PNX diagnosis (0.87 vs 0.46) and equal specificity, 0.99 vs 1.00. LUS is more accurate and faster than chest radiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years in the cardiovascular intensive care unit post cardiac surgery, with a chest tube removed within the past 2 hours.

Exclusion Criteria:

* Patients who were mechanically ventilated or with subcutaneous emphysema due to impaired pleural line visualization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CVICU patients after cardiac surgery
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Pneumothorax | 24 months
  Assess the accuracy of nurse-performed lung ultrasound in the diagnosis of pneumothorax post chest tube removal after cardiac surgery compared to chest x-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Moreno Garijo, MD, Principal Investigator — Sunnybrook Health Science Centre; Azad Mashari, MD, Principal Investigator — University Health Network, Toronto